CLINICAL TRIAL: NCT05434169
Title: Effect of POsitive Therapeutic Communication on PAIN and Anxiety During Arterial Blood Gas Standardized Procedures in the Emergency Department Compared With Traditional Communication: a Monocentric Randomized Controlled Trial
Brief Title: Effect of Positive Therapeutic Communication on Pain
Acronym: POPAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Fribourgeois (Other)
Responsible Party: Principal Investigator, Christophe Le Terrier, Dr., Hôpital Fribourgeois
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2022-00685
Record Dates: First submitted 2022-06-13; First posted 2022-06-27 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Effect of Positive Therapeutic Communication on Pain
Keywords: Pain; Therapeutic communication; Hypnosis; Emergency department; Arterial blood gas; Blood sampling
MeSH Terms: conditions — Pain; Emergencies | interventions — Blood Gas Analysis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Positive Therapeutic communication (Experimental)
  Interventions: Biological: Arterial Blood Gas
- Nocebo communication (Active Comparator)
  Interventions: Biological: Arterial Blood Gas
- Neutral communication (Active Comparator)
  Interventions: Biological: Arterial Blood Gas

INTERVENTIONS:
Biological: Arterial Blood Gas — The procedure of arterial blood collection will be conducted in a seated position for all three groups. The patient is in a supine position, with the forearm comfortably placed on a small table. The needle used for blood collection is a 25 gauge needle without local anesthetic. This method of sampling is identical to the one used in daily practice in the Emergency department of Fribourg

SUMMARY:
Pain, defined as a disagreeable sensory or emotional experience, is the most frequent symptom among patients admitted to the emergency department (ED). It is estimated that this symptom can be observed in almost 80% of patients upon their arrival to the ED. Despite several international recommendations concerning pain management, pain in the context of an emergency situation often remains underestimated. Medical procedures, such as venous or arterial blood collection, which are essential for diagnostic management and patient care, can also generate pain and a high level of stress for patients who are already weakened by their underlying condition. This is known as "care-related pain".

Arterial blood gas (ABG) sampling is necessary to assess the gravity of the patient's condition and is a procedure conducted routinely in the ED. In a medium-size hospital (30,000 hospitalizations per year), approximately 1000 ABG tests are conducted annually. However, ABG collection is generally associated with pain and patient anxiety.

In order to decrease the perception of pain linked to the collection of arterial blood, several methods have been studied, such as applying a topical anesthetic cream (lidocaine, xylocaine) or a subcutaneous infection of lidocaine prior to the procedure. Given that ABG collection is often performed in emergency situations and that the anesthetic cream must be applied at least one hour before sampling, this method is not adapted to emergency practices. In a previous study, a subcutaneous injection of lidocaine did not allow to significantly reduce pain during radial artery puncture. Similarly, another study using ultrasound guidance for ABG sampling did not show any significant decrease in pain, the rate of immediate complications, or physician satisfaction.

Apart from the therapeutic tools commonly used, communication is a key element of care. In routine practice, caregivers inform patients that they are going to perform a potentially painful act. However, forewarning a patient that one will perform a painful act increases the perception of pain. It has also been shown that a communication strategy including the use of positive, kind or reassuring terms ("let me reassure you…", "are you comfortable?", "are you warm enough?") can contribute to decreasing the pain, while conversely, the choice of terms with a negative connotation ("okay, this might sting", "don't panic", "are you in pain?", "are you cold?") may increase the perception of pain and provoke a sense of discomfort. In the latter case, this is known as the "nocebo" effect. A communication strategy including reassuring terms, perceived by the brain as an agreeable information, allows to decrease the penibility dimension or connotes otherwise the pain in order to make it more bearable, thus modulating the painful perception. The objective of this strategy is that the painful message becomes less present as much as possible and that the patient benefits from a feeling of control. This procedure is widely used in hypnosis communication and is based on a neurobiological rationale, i.e., an increase in the secretion of endogenous opioids affecting the pain modulation networks decreases transmission in the pain pathways, thus leading to a release of dopamine in the striatum. This technique has already shown to be of benefit in patient management in various domains, such as anesthesia and pediatrics.

Arrival at the ED can induce a particular state of consciousness linked to anxiety and a heightened suggestibility of negative communication. Although several studies have compared the impact of verbal attitudes, notably in the domain of anesthesia and mainly with staff already trained in hypnosis, to our knowledge, none has studied the effect of positive communication by caregivers or physicians among a patient population in the ED setting. Given the limited therapeutic options to relieve the pain and discomfort of blood collection performed in the ED, we would like to evaluate in this study the potential benefit of positive therapeutic communication on pain and anxiety among patients who require ABG compared to nocebo or neutral communication.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Patients scheduled to undergo radial ABG collection during their visit to the ED to allow to pursue routine care.
* Free and informed consent of the patient received orally from one of the study investigators at study entry.

Exclusion Criteria:

* Vital emergency requiring immediate resuscitation
* Patients incapable of judgement.
* Patients with conditions that render them unable to participate in the intervention of the present study, e.g., cognitive impairment, major hearing loss without the use of hearing aids, acute psychiatric disorders, under intravenous or oral sedation.
* Patients with an insufficient understanding of the French language as defined by self-evaluation.
* Local anesthesia (subcutaneous, transdermal patch) at the point of ABG puncture.
* Patients already treated with anxiolytics or sedatives during care at the ED.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-28 (Actual)

PRIMARY OUTCOMES:
Change of Pain | Change of Pain at 3 minutes after the procedure from baseline
  Self-evaluation of maximum pain felt by the patient during collection of an ABG sample on a Verbal Rating Scale (VRS) (0 = no pain - 10 = worst imaginable pain)

SECONDARY OUTCOMES:
Change of Comfort | Change of Comfort at 3 minutes after the procedure from baseline
  Self-evaluation of patient comfort using a simple comfort VRS (0 = no comfort - 10 = most comfortable imaginable)
Change of Anxiety | Change of Anxiety at 3 minutes after the procedure from baseline
  Self-evaluation of patient anxiety using a simple anxiety VRS (0 = no anxiety - 10 = the worst anxiety imaginable)
Puncture failure | at 3 minutes after the procedure
  The success of the first arterial puncture will be assessed by the accredited evaluator at the end of the procedure by the number of puncture points visible on the patient's skin. Possible response: one puncture visible, yes/no.
Global satisfaction with the communication strategy used | at 3 minutes after the procedure
  Evaluation by the patient at the end of the procedure using a numeric scale of 0 to 10 (0 = extremely dissatisfied - 10 = extremely satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Firbourg Hospital, Fribourg, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schmutz T, Le Terrier C, Ribordy V, Iglesias K, Guechi Y. The Effect of Positive Therapeutic Communication on Pain (POPAIN) and Anxiety During Arterial Blood Gas Standardized Procedures in the Emergency Department Compared to Traditional Communication: Protocol for a Monocentric Randomized Controlled Trial. JMIR Res Protoc. 2023 Jun 13;12:e42043. doi: 10.2196/42043. PMID 37310776